CLINICAL TRIAL: NCT03817619
Title: Bioequivalence Study of CRUshed ElbaSvir/GrAzoprevir compareD to the wholE Tablet (CRUSADE-2)/Hep-NED005
Brief Title: Bioequivalence Study of Crushed Elbasvir/Grazoprevir Compared to the Whole Tablet
Acronym: CRUSADE-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF 17.01
Record Dates: First submitted 2019-01-21; First posted 2019-01-25 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis C; Deglutition Disorders
MeSH Terms: conditions — Hepatitis C; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Open-label, 2-period, randomised, cross-over, single-centre, phase I, single-dose trial in 14 healthy adult subjects.
  Intrasubject comparison of PK parameters after different administrations of Zepatier
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment R (reference) (Active Comparator): Single-dose ELB/GZR as a whole tablet in a fasted state.
  Interventions: Drug: Zepatier whole tablet
- Treatment T (test) (Experimental): Single-dose crushed ELB/GZR in a fasted state.
  Interventions: Drug: Zepatier crushed tablet

INTERVENTIONS:
Drug: Zepatier whole tablet — Single-dose ELB/GZR as a whole tablet in a fasted state.
  Arms: Treatment R (reference)
Drug: Zepatier crushed tablet — Single-dose crushed ELB/GZR in a fasted state.
  Arms: Treatment T (test)

SUMMARY:
Elbasvir/grazoprevir (Zepatier®) is a once-daily tablet for the treatment of chronic hepatitis C virus (HCV) GT1a, 1b or 4 infection containing the NS5A inhibitor elbasvir (ELB) 50 mg and the NS3/4A protease inhibitor grazoprevir (GZR) 100 mg.

For patients with swallowing difficulties, administration of whole tablets can be problematic. In addition, HCV patients that are hospitalized (at intensive care units) due to severe illness (co-infections/ liver failure) might not be able to swallow medication. Therefore it is useful to know whether it is possible to administer ELB/GZR through a different route, like a feeding tube.

In daily practice, information about the safety and efficacy of crushed tablets is lacking which might result in noncompliance, interruption or discontinuation of expensive HCV therapy. However, it is not recommended to interrupt treatment because there is no evidence about the efficacy of the therapy after discontinuation (and restarting).

Currently, patients and healthcare professionals are crushing tablets without information about efficacy and safety. Depending on the biopharmaceutical characteristics of a drug formulation, crushing tablets can lead to altered pharmacokinetics of drugs.

It is important to know whether pharmacokinetic parameters are influenced by crushing of tablets; both a decrease and an increase in exposure may occur. A decrease of the plasma concentrations of ELB and/or GZR potentially reduces the therapeutic effect of the drugs. Higher doses or switching to other HCV-drugs might be needed. In contrast, in case a higher Cmax and/or AUC occurs there might be an increased risk of toxicity.

As a result, crushing the drug is a contra-indication based on the available data. Therefore this study will be conducted to investigate whether a crushed ELB/GZR tablet is bioequivalent to ELB/GZR as a whole tablet.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 and not older than 55 years at screening.
* Subject does not smoke more than 10 cigarettes, 2 cigars, or 2 pipes per day for at least 3 months prior to Day 1.
* Subject weighs at least 40 kg.
* Subject has a Quetelet Index (Body Mass Index) of 18 to 30 kg/m2, extremes included.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* Subject is in good age-appropriate health condition as established by medical history, physical examination, and electrocardiography, results of biochemistry, hematology and urinalysis testing within 4 weeks prior to Day 1. Results of biochemistry, hematology and urinalysis testing should be within the laboratory's reference ranges. If laboratory results are not within the reference ranges, the subject is included on condition that the Investigator judges that the deviations are not clinically relevant. This should be clearly recorded.
* Subject has a normal blood pressure and pulse rate, according to the Investigator's judgment.

Exclusion Criteria:

* Creatinine clearance below 60 mL/min.
* Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
* Positive hepatitis B or C test
* Pregnant female (as confirmed by an hCG test performed less than 4 weeks before day 1) or breast-feeding female. Female subjects of childbearing potential without adequate contra-ception, e.g. hysterectomy, bilateral tubal ligation, (non-hormonal) intrauterine device, total abstinence, double barrier methods, or two years post-menopausal. They must agree to take precautions in order to prevent a pregnancy throughout the entire conduct of the study.
* Therapy with any drug (for two weeks preceding Day 1), except for acetaminophen (max 2 gram/day).
* Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), psychiatric disorders, gastro-intestinal disorders, renal and hepatic disorders (clinically relevant increased ALAT/ASAT or hyperbilirubinemia), hormonal disorders (especially diabetes mellitus), coagulation disorders.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* History of or current abuse of drugs, alcohol or solvents (positive drugs of abuse test).
* Inability to understand the nature and extent of the study and the procedures required.
* Participation in a drug study within 60 days prior to Day 1.
* Donation of blood within 60 days prior to Day 1.
* Febrile illness within 3 days before Day 1.
* Co-worker of Radboud university medical center.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Bioequivalence AUC0-72h | 72 hours
  Determination of elbasvir/grazoprevir AUC0-72h by noncompartmental analysis. Descriptive statistics for the plasma concentrations of elbasvir/grazoprevir at each sampling time. Descriptive statistics for each PK parameter per treatment (geometric mean + CV%).
  Geometric Mean Ratios and 90% confidence intervals of pharmacokinetic parameters of treatment T (Test) vs. treatment R (Reference). AUC0-72h geometric mean ratios for elbasvir and grazoprevir with a 90% Cl falling entirely within the range of 0.7 to 1.43 are considered bioequivalent.

SECONDARY OUTCOMES:
Bioequivalence (Cmax) | 18 days
  Determination of grazoprevir Cmax by noncompartmental analysis. Geometric Mean Ratios and 90% confidence intervals of pharmacokinetic parameters of T (Test) vs. R (Reference).
  Cmax geometric mean ratios for elbasvir and grazoprevir with a 90% Cl falling entirely within the range of 0.7 to 1.43 are considered bioequivalent.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | 18 days
  Adverse events after intake of elbasvir/grazoprevir tablets in healthy adult volunteers.

CONTACTS AND LOCATIONS:
Locations (1):
- RTCCS Radboudumc, Nijmegen, Netherlands

REFERENCES:
- [Background] Pijnenburg DWM, van Seyen M, Abbink EJ, Colbers A, Drenth JPH, Burger DM. Pharmacokinetic similarity demonstrated after crushing of the elbasvir/grazoprevir fixed-dose combination tablet for HCV infection. J Antimicrob Chemother. 2020 Sep 1;75(9):2661-2665. doi: 10.1093/jac/dkaa230. PMID 32544221
- See also: paper — https://pubmed.ncbi.nlm.nih.gov/32544221/